CLINICAL TRIAL: NCT00732420
Title: A Phase I Open-label Study of the Safety, Tolerability, and Pharmacokinetics of Two Schedules of Oral Topotecan in Combination With Pazopanib in Subjects With Advanced Solid Tumors
Brief Title: Open-label Study of Topotecan and Pazopanib in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HYT109091
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumours
Keywords: pazopanib; Phase I; topotecan; Advanced Solid Tumors
MeSH Terms: interventions — Topotecan; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A (Experimental): Daily oral pazopanib in combination with weekly oral topotecan. Initially rising dose to determine the maximum tolerated dose: finally an expanded cohort treated at the maximum tolerated dose.
  Interventions: Drug: topotecan; Drug: pazopanib
- Treatment Arm B (Experimental): Daily oral pazopanib in combination with oral topotecan given for 5 consecutive days every 21 days. Initially rising dose to determine the maximum tolerated dose; finally an additional cohort of patients treated at the maximum tolerated dose.
  Interventions: Drug: topotecan; Drug: pazopanib

INTERVENTIONS:
Drug: topotecan — Topoisomerase I inhibition.
Drug: pazopanib — Tyrosine kinase inhibitor

SUMMARY:
To determined what dose of topotecan can be safely given with daily pazopanib.

DETAILED DESCRIPTION:
A Phase I Open-label Study of the Safety, Tolerability, and Pharmacokinetics of Two Schedules of Oral Topotecan in combination with Pazopanib in Subjects with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria -

* signed, written informed consent.
* at least 18 years of age.
* ECOG performance status 0 or 1.
* Subjects must have histologically or cytologically confirmed diagnosis of advanced cancer and a solid tumor malignancy that has relapsed or is refractory to standard therapy or for which there is no established therapy.
* able to swallow and retain oral medications.
* females are eligible to enter and participate in this study providing adequate established contraception is being practiced.

Exclusion Criteria

* had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* received an investigational drug within 30 days or 5 half-lives (whichever is longer).
* received prior treatment with pazopanib/investigational anti-angiogenic compounds.
* presence of uncontrolled infection.
* pregnant or lactating.
* poorly controlled hypertension (SBP of ? 140 mmHg, or DBP of ? 90 mmHg.
* Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.-
* arterial thrombi, myocardial infarction, admission for unstable angina, uncontrolled or symptomatic arrhythmia, cardiac angioplasty, or stenting within the last 6 months.
* any unresolved bowel obstruction or diarrhea ? Grade 1.
* received an allogeneic bone marrow transplant.
* known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or topotecan.
* any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the study.
* psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* clinical history, current alcohol or illicit drug use which, in the judgment of the investigator, would interfere with the subject's ability to comply with the dosing schedule and protocol-specified evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-09-24 (Actual); Primary Completion 2013-06-12 (Actual); Study Completion 2013-06-12 (Actual)

PRIMARY OUTCOMES:
First course tolerability with rising dose of topotecan to determine the maximum tolerated dose of topotecan when given with pazopanib daily. | 5 weeks

SECONDARY OUTCOMES:
Indications of efficacy through tumour shrinkage. Specific biomarker analysis. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Philadelphia, Pennsylvania, United States
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Utrecht

REFERENCES:
- See also: Results for study HYT109091 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/HYT109091?search=study&study_ids=HYT109091#rs